CLINICAL TRIAL: NCT05011461
Title: The Effect of Topical Almond Oil vs. Topical Retinol on The Appearance of Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Raja Sivamani, MD, Associate Professor of Clinical Dermatology, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1666459
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Wrinkles; Skin
MeSH Terms: interventions — almond oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond Oil (Experimental): Almond Oil Pressed Cold
  Interventions: Other: Almond Oil
- Topical Retinol (Active Comparator): Retinol Lotion 0.5%
  Interventions: Other: Almond Oil

INTERVENTIONS:
Other: Almond Oil — Almond Oil Pressed Cold

SUMMARY:
The purpose of this experiment is to analyze wrinkle severity, the skin barrier and facial pigmentation level after topical almond oil application, compared to the use of topical retinol. Both the almond oil and the 0.5% topical retinol studied is investigational.

DETAILED DESCRIPTION:
The natural cosmetic market is a multi-billion-dollar industry. Nutraceuticals and foodbased cosmetics are a growing trend within dermatology. Almonds are a rich dietary source of a range of fatty acids, phytochemical polyphenols, and antioxidants [1]. The previous study done by Dr. Raja Sivamani was a double blinded study that compared oral almond intake to a calorie matched non-nut-based intake over 12 weeks.The study determined that that there was a statistically significant improvement in wrinkle severity and pigment intensity in the women that received almond supplementation. This proposal aims to now understand how the topical application of almond oil may influence the appearance of wrinkles and facial tone in post-menopausal women. Almond oil is rich in fatty acids and alpha-tocopherol [2]. Tocopherol inhibits melanogenesis in melanocytes [3] and topical alpha tocopherol has been shown to improve skin antioxidants and hyperpigmentation [4, 5].

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women of Fitzpatrick skin types 1 and 2

Exclusion Criteria:

* Those with a nut allergy
* Smoking is an independent risk factor and serves as a confounder for the development of facial wrinkles and photoaging [14]. Therefore, current smokers, those that have smoked within the past year, and former smokers with greater than a 20-pack year history of smoking will be excluded.
* Those with an autoimmune photosensitive condition or a known genetic condition with a deficiency in collagen production (such as Ehlers-Danlos syndromes) will be excluded as this can be a confounder for facial wrinkles.
* Those who have undergone any cosmetic procedures to the face in the 4 months prior to enrollment in the opinion of the investigator. People that have undergone deeper chemical peels (TCA based peels) within 1 year prior to enrollment will also not be eligible.
* Individuals who are unwilling to discontinue vitamin E food sources during the washout and intervention. This includes

  * Vitamin E containing supplements.
  * Sunflower seeds or sunflower oil.
  * All nuts.
* Individual who are unwilling to discontinue topical cosmetic products during the duration of the study or unwilling to undergo a 2-week washout of topicals that are known to modulate collagen and pigment:

  * Retinoids such as tretinoin, adapalene, retinol, except as provided by the study.
  * Antioxidant ingredients such as vitamin C or vitamin E.
  * Pigment reducing agents such as hydroquinone, a retinoid, azelaic acid, kojic acid, pomegranate seed oil, and other similar agents per the discretion of the investigator, except for the retinol that is provided in this study.
  * Topicals that contain a nut oil or nut extract as part of their ingredient list.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Appearance of wrinkle severity | 12-weeks
  Facial wrinkles will be assessed with the use of a validated high resolution facial modeling system. The high-resolution facial modeling system will be performed with the 3D Clarity Pro® Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA) and will specifically assess for wrinkle severity and wrinkle length as was performed in the previous pilot study.

SECONDARY OUTCOMES:
Appearance of facial color tone and evenness | 12-weeks
  The facial color tone and evenness will be measured with a SkinColor Catch from Delfin Technologies. This device shows the RGB Colors, CIE L*a*b* and L*c*h* color space coordinates when the devivce is applied to the skin. Included is the link to the device (http://www.truesystem.co.kr/product/pdf/SkinColorCatch%20Brochure%202016.pdf).
Appearance of facial redness | 12-weeks
  We will quantify the presence of facial redness with a SkinColor Catch from Delfin Technologies. We will measure the RGB colors and average them from each participant for each of the visits. Skin pigment, including the presence of redness, will be measured using a SkinColorCatch from Delfin Technologies . This device shows the RGB Colors, CIE L*a*b* and L*c*h* color space coordinates when the devivce is applied to the skin. Included is the link to the device (http://www.truesystem.co.kr/product/pdf/SkinColorCatch%20Brochure%202016.pdf).
Subjective tolerability | 12-weeks
  To assess tolerability, we are going to use a Tolerability Assessment Questionnaire. The patient fills out the questionnaire on whether they currently have or had any itching, burning, stining, scaling, erythema, hypopigmentation or hyperpigmentation during application of the product. They measure any of the symptoms on a scale of 0-3, 0 being none, 3 being severe. They can also hand write any other effects that they noticed from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, M.D., Principal Investigator — UC Davis Dermatology
Locations (1):
- UC Davis Department of Dermatology, Clinical Trials Unit, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No